CLINICAL TRIAL: NCT02203682
Title: The Effect of Subantimicrobial Dose Doxycycline in Mild Thyroid-Associated Ophthalmopathy
Brief Title: Doxycycline Treatment in Mild Thyroid-Associated Ophthalmopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013MEKY033
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Graves Ophthalmopathy; Graves Disease; Thyroid-associated Ophthalmopathy; Thyroid Diseases; Endocrine System Diseases; Eye Diseases, Hereditary; Hyperthyroidism; Autoimmune Diseases; Immune System Diseases
Keywords: Graves' orbitopathy; Graves´ ophthalmopathy; Thyroid eye disease; Thyroid-associated ophthalmopathy; Doxycycline; EUGOGO; CAS
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Thyroid Diseases; Endocrine System Diseases; Eye Diseases, Hereditary; Hyperthyroidism; Autoimmune Diseases; Immune System Diseases | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Experimental): Tablets Doxycycline 50 mg PO per day for 12 weeks
  Interventions: Drug: Doxycycline hyclate
- Placebo (Placebo Comparator): Tablet placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline hyclate — Tab. Doxycycline 50 mg PO per day for 12 weeks
  Arms: Doxycycline
Drug: Placebo — Tablet placebo for 12 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects of subantimicrobial dose doxycycline (50 mg/d), administered for 12 weeks, on patients with mild Thyroid-Associated Ophthalmopathy (TAO).

DETAILED DESCRIPTION:
Thyroid-Associated Ophthalmopathy is an autoimmune disease that can be treated by corticosteroids and surgery. But they often cause severe side-effects and are usually used for treating moderate-sever and sight-threatening TAO. Wait and see will be the first choice for the patient with mild TAO.

Subantimicrobial dose (SD) doxycycline displays a strong anti-inflammatory and immunomodulatory function, which is independent of its antibiotic properties. Data from clinical trials demonstrated that SD doxycycline was effective in moderating inflammation in a variety of autoimmune diseases, such as rheumatoid arthritis, multiple sclerosis, rosacea and periodontitis.

We propose to test the effect of subantimicrobial dose doxycycline for mild TAO.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Thyroid-associated ophthalmopathy
* Mild TAO
* Normal serum free thyroxine and free triiodothyronine concentrations
* No previous specific therapy for TAO, except for local measures
* Written informed consent is obtained

Exclusion Criteria:

* Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing, or lactating females
* Uncontrolled diabetes or hypertension
* History of mental / psychiatric disorder
* Hepatic dysfunction (Alb, AST, ALT and Alkaline phosphates levels must be within normal range for eligibility)
* Renal impairment (Urea and Creatinine levels must be within normal range)
* Tetracycline allergy or intolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
the rate of improvement | 12 weeks
  Improvement was defined that at least one item was met in the study eye without deterioration in any item of both eyes:
  1. reduction of eyelid aperture by at least 2mm;
  2. reduction in exophthalmos by at least 2mm;
  3. increase in ocular motility by at least 8 degrees in any duction;
  4. increase on either GO-QOL scales by at least 6 points. The higher of the rate of improvement gets, the better the outcome is. The primary outcome ranges from -100% to 100%.

SECONDARY OUTCOMES:
Clinical Activity Score (CAS) | 4weeks and 12 weeks
  Patients will be assessed according to the 7 item European Group on Graves' Ophthalmopathy (EUGOGO) amended Clinical Activity Score (CAS) For each item present, one point is given. The sum of the points is the total score ranges from 0 to 7.
  1. Spontaneous orbital pain.
  2. Gaze evoked orbital pain.
  3. Eyelid swelling that is considered to be due to active (inflammatory phase) GO.
  4. Eyelid erythema.
  5. Conjunctival redness that is considered to be due to active (inflammatory phase) GO (ignore "equivocal" redness).
  6. Chemosis.
  7. Inflammation of caruncle or plica.
Proptosis measured by Hertel instrument | 4weeks and 12 weeks
  For the assessment of proptosis, the same Hertel instrument and ideally the same observer should be used on each occasion. Additionally the same intercanthal distance (ICD) should be used on each occasion. The Hertel values will be measured for each eye at each visit and repeated three times. The mean value is recorded. Proptosis ranges from 10mm to 30mm.
Eyelid aperture | 4weeks and 12 weeks
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. These measurements are repeated three times, and the mean value is recorded. When performed this assessment, participants should relax their eyes and keep looking ahead and the observers should keep the ruler perpendicular to their eyelid.
Lid retraction | 4weeks and 12 weeks
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. The upper eyelid positions above (positive value) and below (negative value) the superior limbus and The lower eyelid positions above (positive value) and below (negative value) the posterior limbus were measured in millimeters in primary position. These measurements are repeated three times, and the mean value is recorded.
Lid lag | 4weeks and 12 weeks
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. Lid lag is defined that the lid margin distance in downgaze. The upper eyelid positions above (positive value) and below (negative value) the superior limbus were measured in millimeters.
Eye motility | 4weeks and 12 weeks
  The head of each participant is adjusted to fix on the modified perimeter to set the visual axis of the examined eye on the center of the optimal visual target in visual chart. The other eye should be covered. The examined eye should follow the movement of the visual target until the participant cannot identify the exact visual target in vertical and horizontal directions. And the extreme scales of these four directions are obtained. These measurements are repeated three times, and the mean value is recorded.
Graves' Ophthalmopathy Quality of Life Scale | 4weeks and 12 weeks
  The Graves' Ophthalmopathy Quality of Life (GO-QOL) questionnaire (Terwee & al, 1998) includes visual functioning and psychosocial functioning. A raw score of each part is calculated by adding each score of 8 question, namely 1, 2, or 3 for each question which means marked, mild, or absent limitation, the final score ranging from 0 (full limitation) to 100 (no limitation) is calculated as the following rule: (raw score - 8) ÷ 16 × 100]. GO-QOL will be completed at screening, weeks 0, 4, 12. were also recorded to assess activity of TAO and impact on quality of life respectively.
  The GO-QOL is a 16 item self-administered questionnaire used to assess the perceived effects of TAO by the patients on their daily physical and psychosocial functioning.
C-OSDI | 4weeks and 12 weeks
  The Ocular Surface Disease Index (OSDI), developed by the Outcomes Research Group at Allergan Inc (Irvine, Calif), is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation and vision-related functioning.
the category of adverse events and the frequency of the occurrence of adverse events | 4weeks and 12 weeks
  The category of adverse events and the frequency of the occurrence of adverse events are listed to describe the safety.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Principal Investigator — Zhongsh Ophthalmic Center
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Pan Y, Chen YX, Zhang J, Lin ML, Liu GM, Xu XL, Fan XQ, Zhong Y, Li Q, Ai SM, Xu W, Tan J, Zhou HF, Xu DD, Zhang HY, Xu B, Wang S, Ma JJ, Zhang S, Gan LY, Cui JT, Li L, Xie YY, Guo X, Pan-Doh N, Zhu ZT, Lu Y, Shi YX, Xia YW, Li ZY, Liang D. Doxycycline vs Placebo at 12 Weeks in Patients With Mild Thyroid-Associated Ophthalmopathy: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 Nov 1;140(11):1076-1083. doi: 10.1001/jamaophthalmol.2022.3779. PMID 36173609